CLINICAL TRIAL: NCT06339593
Title: Regional Monitoring of CF Lung Disease After Changes in Mechanical Airway-clearance Treatment
Brief Title: Regional Monitoring of CF Lung Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Jason Woods, PhD, Director, Center for Pulmonary Medicine Imaging Research, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0391
Record Dates: First submitted 2024-02-06; First posted 2024-04-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CF pts on MACT (Other): Males and females from 12 to 21 years old who have been prescribed Mechanical Airway Clearance Therapy for CF.
  Interventions: Drug: Hyperpolarized Xe129
- Self withdrawn ACT (Other): To perform a stepwise ACT re-initiation trial in fifteen 12-21 y.o. patients who have self-withdrawn airway clearance treatment (defined as ≤ 3x/week). UTE and Xe MRI, spirometry, and multiple-breath washout will be performed at baseline, after increasing treatment to 7x/week for 1 week and then 14x/week for 2 weeks, with daily logging to aid compliance and study engagement.
  Interventions: Procedure: Airway-clearance vest; Drug: Hyperpolarized Xe129
- Low MRI abnormalities and high FEV1 (Other): To perform a stepwise ACT withdrawal trial in fifteen 12-21 y.o. patients who have low MRI abnormalities and high FEV1. Patients will be studied at baseline, after decreasing ACT to 7x/week for 1 week, and after decreasing ACT to 3x/week for 1 week.
  Interventions: Procedure: Airway-clearance vest; Drug: Hyperpolarized Xe129

INTERVENTIONS:
Procedure: Airway-clearance vest — Airway clearance devices will be re-initiated for those who have self withdrawn and will be withdrawn temporarily for those who are using them regularly and have high FEV1 and low Xe MRI ventilation defects.
  Arms: Low MRI abnormalities and high FEV1; Self withdrawn ACT
Drug: Hyperpolarized Xe129 — Hyperpolarized Xe MRI is FDA Approved for evaluation of ventilation in adults and children 12 and above and will be used as a diagnostic test here. Earlier studies using Xe MRI have shown its efficacy in exploring CF and other lung diseases in pediatric and adult populations, and it has been found to be much more sensitive to early lung disease than traditional metrics like spirometry and MBW.

SUMMARY:
The main reason for this research study is to learn more about some new tests that are being developing for patients with Cystic Fibrosis (CF) to measure changes in the lungs. In this study, the focus will be to learn how stopping Airway Clearance (ACT) and re-starting ACT can affect these tests. These new tests include using a breathable gas called Xenon (Xe) with MRI (magnetic resonance imaging) to improve the pictures of changes in the lungs. The Xenon (Xe) gas that has been treated to have a larger MRI signal (also called hyperpolarized). The other new test is called LCI (Lung Clearance Index) that can measure how well the lungs are working. The MRI machine used in this study has been approved by the U.S. Food and Drug Administration (FDA) and is commercially available for sale in the USA. Hyperpolarized Xe gas is an FDA-approved, inhaled contrast agent for lung ventilation MRI. The new Xe MRI techniques that are being developed and used for this research study are investigational, meaning these new Xe MRI techniques are not FDA approved, but they are similar to FDA-approved techniques that are used clinically at Cincinnati Children's Hospital Medical Center (CCHMC). Xe gas and the new MRI techniques used in this research study have been used for many years in research, including in many research studies conducted at CCHMC like this one.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a progressive, systemic disease affecting an estimated 30,000 children and adults in the United States (70,000+ worldwide) and is caused by mutations in the gene that encodes the cystic fibrosis transmembrane conductance regulator (CFTR) protein--a chloride and bicarbonate channel that regulates ion transport and mucus composition in CF-affected tissues, such as the lung. In airways this leads to mucus stasis, infection, inflammation, and remodeling that result in mucus plugs, regional lung obstruction, and progressive airway destruction and bronchiectasis. Highly-effective CFTR modulators, which are recently available to >90% of patients, have revolutionized CF clinical care, with large increases in pulmonary function as a result of more effective mucociliary clearance. As a result, burdensome maintenance therapies like mechanical airway clearance treatment (ACT), requiring nearly 2 dedicated hours per day, have been questioned by patients, families, and medical providers. In a recent survey of CF community members, ACT was ranked as the most burdensome chronic therapy, yet is the least studied. Prospective studies of maintenance-therapy withdrawal pose potential ethical risks, since traditional testing via spirometry and/or multiple-breath washout is relatively insensitive to small or regional changes and long-term lung-function reductions often have permanent consequences. Nevertheless, many patients have withdrawn these maintenance therapies against advice from their providers. A major gap in CF management is our ability to monitor lung function sensitively and rapidly as a result of treatment changes, such as partial withdrawal of ACT.

Breakthroughs in structural and functional magnetic resonance imaging (MRI) have demonstrated exquisite sensitivity to regional CF lung disease and can monitor regional and subtle changes over time, without ionizing radiation, even in patients with normal spirometry. As demonstrated in the previous R01 that ultrashort echo time (UTE) MRI provides structural images that rival computered tomography (CT) imaging, with sensitivity to detect all of the structural hallmarks of treatable (e.g., mucus plugs) and permanent lung disease (e.g., bronchiectasis). It has been demonstrated that hyperpolarized 129Xe MRI is more sensitive than any other technique at detecting changes in regional pulmonary ventilation and gas exchange. For the first time, a single modality (MRI) is available to safely monitor regional lung disease and treatment changes before FEV1 declines become permanent. This is a unique opportunity to safely evaluate ACT in CF populations that remain at risk of long-term lung function decline.

ELIGIBILITY:
Inclusion Criteria:

* 1 Written informed consent (and assent when applicable) obtained from subject or subject's legal representative.

  2 Use of highly effective modulators for more than 30 days (ie. Trikafta) 3 Willingness and ability to adhere to the study visit schedule and other protocol requirements.

  4 Documentation of a CF diagnosis with prescription of Mechanical ACT 5 Ages 12-21 inclusive, at the time of consent. 6 Clinically stable with no respiratory tract infection or recent exacerbations. 7 Treating CF physician agreeable to study procedures. Only applicable to Aim 3.

  8 No change in chronic maintenance therapies in the 28 days prior to enrollment.

  9 Ability to cooperate with MRI procedures.

Exclusion Criteria:

1. Standard MRI exclusions (metal implants, claustrophobia).
2. For females of childbearing potential: Positive urine pregnancy test or Lactating.
3. Acute respiratory symptoms (e.g., wheezing) at the time of the MRI
4. Chronic lung or liver or pancreatic disease not related to CF.
5. Any other condition that, in the opinion of the Investigator, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Assessing functional lung abnormalities via Xenon MRI | two weeks
  We will be using Hyperpolarized Xenon MRI images of participants with Cystic Fibrosis

SECONDARY OUTCOMES:
Assessing patients who have self-withdrawn airway clearance treatment to determine ventilation abnormalities. | two weeks
  UTI MRI will be used to measure participants airway clearance
Assessing patients who have self-withdrawn airway clearance treatment to determine ventilation abnormalities. | two weeks
  Spirometry will be used to measure participants airway clearance
Assessing patients who have self-withdrawn airway clearance treatment to determine | 2 weeks
  Multiple-breath washout will be used to measure participants airway clearance

OTHER OUTCOMES:
Change in Xenon Ventilation Defect Process (VDP) | 4 weeks
  Examination of the lung function decline of patients after airway clearance techniques (ACT) withdrawal. The baseline visit will be measured with UTE.
Change in Xenon Ventilation Defect Process (VDP) | 4 weeks
  Examination of the lung function decline of patients after airway clearance techniques (ACT) withdrawal. The baseline visit will be measured with Xenon MRI.
Changes in Xenon Ventilation Defect Process (VDP) | 4 weeks
  Examination of the lung function decline of patients after airway clearance techniques (ACT) withdrawal. The baseline visit will be measured with Spirometry.
Changes in Xenon Ventilation Defect Process (VDP) | 4 weeks
  Examination of the lung function decline of patients after airway clearance techniques (ACT) withdrawal. The baseline visit will be measured with Lung Clearance Index (LCI).

CONTACTS AND LOCATIONS:
Overall Officials: Jason C Woods, PhD, Principal Investigator — Cincinnati Children's Hospital Medica Center
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No